CLINICAL TRIAL: NCT03559101
Title: Characterization of the Effects of Amino Acid/Electrolyte-based Beverages on Hydration Status in Young and Older Subjects
Brief Title: Effects of Amino Acid/Electrolyte-based Beverages on Hydration Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W. Larry Kenney (Other)
Responsible Party: Sponsor-Investigator, W. Larry Kenney, Professor of Physiology and Kinesiology, Penn State University
Organization: Penn State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY6412
Record Dates: First submitted 2018-05-22; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Dehydration
Keywords: Hydration; Plasma Volume; Amino acids; Glucose; Electrolytes; Fluid Retention; Aging; Beverage Hydration Index; Dehydration; Oral Rehydration
MeSH Terms: conditions — Dehydration | interventions — gatorade

STUDY DESIGN:
Intervention Model Description: Two groups of subjects (young, older) participate in five experiments, one for each of five beverage pretreatments. Pretreatments are consumed immediately prior to the experiment. The experiments are conducted in randomized order. The trials are identical and separated by at least five days.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The ingredients-list is masked on the bottles of beverage. Test beverages are coded. The research nurse logs the code, administers the test beverage, and discards the empty bottle prior to the experiment and in the absence of the investigator and outcomes assessor. The investigator and outcomes assessor do not have access to the log. Subjects do not discuss the beverages with the investigator and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Beverage 1 - Control (Active Comparator): Distilled Water
  Interventions: Other: Distilled water
- Beverage 2 (Experimental): Medical Food 1 (8 amino acids, 60 mmol/L Na, 20 mmol/L K + citrate, Cl)
  Interventions: Other: Medical Food 1
- Beverage 3 (Experimental): Medical Food 2 (8 amino acids, 30 mmol/L Na, 10 mmol/L K + citrate, Cl)
  Interventions: Other: Medical Food 2
- Beverage 4 (Experimental): Pedialyte
  Interventions: Other: Pedialyte
- Beverage 5 (Experimental): Gatorade
  Interventions: Other: Gatorade

INTERVENTIONS:
Other: Distilled water — Commercially available beverage
  Subjects collect all morning urine and drink 500 milliliters of water. Baseline vital measurements (heart rate, blood pressure, oral temperature) and body weight collected Baseline blood samples and urine collected Beverage pretreatment consumed (1 liter over 30 minutes) Body weight measured and blood and urine collected at 5 minutes, 10 minutes, 15 minutes, and then every 30 minutes for 4 hours post beverage consumption
  Arms: Beverage 1 - Control
Other: Medical Food 1 — Commercially available beverage
  Subjects collect all morning urine and drink 500 milliliters of water. Baseline vital measurements (heart rate, blood pressure, oral temperature) and body weight collected Baseline blood samples and urine collected Beverage pretreatment consumed (1 liter over 30 minutes) Body weight measured and blood and urine collected at 5 minutes, 10 minutes, 15 minutes, and then every 30 minutes for 4 hours post beverage consumption
  Arms: Beverage 2
Other: Medical Food 2 — Commercially available beverage
  Subjects collect all morning urine and drink 500 milliliters of water. Baseline vital measurements (heart rate, blood pressure, oral temperature) and body weight collected Baseline blood samples and urine collected Beverage pretreatment consumed (1 liter over 30 minutes) Body weight measured and blood and urine collected at 5 minutes, 10 minutes, 15 minutes, and then every 30 minutes for 4 hours post beverage consumption
  Arms: Beverage 3
Other: Pedialyte — Commercially available beverage
  Subjects collect all morning urine and drink 500 milliliters of water. Baseline vital measurements (heart rate, blood pressure, oral temperature) and body weight collected Baseline blood samples and urine collected Beverage pretreatment consumed (1 liter over 30 minutes) Body weight measured and blood and urine collected at 5 minutes, 10 minutes, 15 minutes, and then every 30 minutes for 4 hours post beverage consumption
  Arms: Beverage 4
Other: Gatorade — Commercially available beverage
  Subjects collect all morning urine and drink 500 milliliters of water. Baseline vital measurements (heart rate, blood pressure, oral temperature) and body weight collected Baseline blood samples and urine collected Beverage pretreatment consumed (1 liter over 30 minutes) Body weight measured and blood and urine collected at 5 minutes, 10 minutes, 15 minutes, and then every 30 minutes for 4 hours post beverage consumption
  Arms: Beverage 5

SUMMARY:
Older adults typically do not drink later in the day to avoid the necessity of interrupting sleep to urinate. Sometimes they also limit ingestion of fluids to avoid the need to urinate when engaged in certain activities such as traveling or attending an event. Therefore, beverages that have greater fluid retention in the body leading to a more sustained positive hydration status could be advantageous in such situations. The composition of a beverage as well as other factors such as volume ingested and metabolism of components can affect the retention of the fluid in the body. Age may be another factor. The beverage hydration index (BHI), first described in 2016, was used to indicate the hydration response to thirteen well-known beverages in young male adults. The current study assesses the BHI of four beverages and how that response is affected by age following the standardized protocol. The four beverages have been chosen for inclusion in this study because they have been used by older adults to prevent dehydration.

DETAILED DESCRIPTION:
Subjects sign an informed consent form and undergo a medical screening prior to participation. The screening includes a physical exam, anthropometry, chemical and lipid profiles, as well as measures of liver and renal function. The subjects are assigned to one of two groups based upon age.

Subjects participate in five experimental trials, one for each of the five beverages. The beverages are commercially-available and contain ingredients that are generally recognized as safe (GRAS). The order of the beverages is randomized. The list of ingredients on the bottle containing the beverage is obscured. The trials are identical and separated by at least five days. For each experiment, baseline measurements are conducted. Then the subjects consume one liter of the test beverage over thirty minutes. Additional measurements are performed thirty minutes post ingestion and then every hour for four hours post ingestion.

This study yields two BHI numbers for each beverage, one number for each study-group. The BHI numbers are indicative of the amount of fluid remaining in the body four hours after consumption of the beverage. The BHI number is inversely related to the amount of urine produced over the four hours. A greater BHI number indicates better fluid retention and maintenance of plasma volume.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years or ≥60 years

Exclusion Criteria:

* cardiovascular, renal, or digestive diseases
* pregnancy
* breastfeeding
* smoking and/or use of nicotine-containing products
* illegal/recreational drug use
* medications that alter fluid balance (e.g., diuretics)
* allergy to Latex
* men with prostate issues that interfere with urination.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Beverage hydration index (BHI) | One BHI for each beverage for each age group is calculated and reported through study completion, an average of 1 year.
  Indicative of amount of fluid remaining in body four hours post consumption of beverage. Inversely related to amount of urine produced over 4 hours. Larger BHI number indicates better fluid retention and maintenance of plasma volume.

SECONDARY OUTCOMES:
Body Mass | Baseline before consumption of beverage and then 5 minutes, 10 minutes, 15 minutes, and then every 30 minutes for 4 hours post beverage consumption
  Body weight measured on scale
Urine Mass | Baseline before consumption of beverage and then 5 minutes, 10 minutes, 15 minutes, and then every 30 minutes for 4 hours post beverage consumption
  Weight of urine produced

CONTACTS AND LOCATIONS:
Overall Officials: William L Kenney, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Clarke MM, Stanhewicz AE, Wolf ST, Cheuvront SN, Kenefick RW, Kenney WL. A randomized trial to assess beverage hydration index in healthy older adults. Am J Clin Nutr. 2019 Jun 1;109(6):1640-1647. doi: 10.1093/ajcn/nqz009. PMID 31051498